CLINICAL TRIAL: NCT01896466
Title: Influence of Neuromodulation on Gait and Balance
Brief Title: Enhanced Gait and Balance Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2013-0394
Record Dates: First submitted 2013-06-10; First posted 2013-07-11 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Aging; Accidental Falls
Keywords: Fall Risk; Gait; Dynamic Balance; Static Balance; Neuromodulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Young Adults - Intervention (Active Comparator): Healthy subjects between the ages of 18-39 will participate in Cranial Nerve Non-Invasive Neuromodulation gait and balance training.
  Interventions: Device: Cranial Nerve Non-Invasive Neuromodulation
- Healthy Older Adults - Control (Active Comparator): Healthy subjects between age 65+ will participate in Sham Cranial Nerve Non-Invasive Neuromodulation gait and balance training.
  Interventions: Behavioral: Sham Cranial Nerve Non-Invasive Neuromodulation
- Healthy Older Adults - Intervention (Active Comparator): Healthy subjects age 65+ will participate in Cranial Nerve Non-Invasive Neuromodulation enhanced gait and balance training.
  Interventions: Device: Cranial Nerve Non-Invasive Neuromodulation
- Older Fallers - Control (Sham Comparator): Subjects who are age 65+ with a history of 1-3 falls in the previous six months will participate in Sham Cranial Nerve Non-Invasive Neuromodulation gait and balance training.
  Interventions: Behavioral: Sham Cranial Nerve Non-Invasive Neuromodulation
- Older Fallers - Intervention (Experimental): Subjects who are age 65+ with a history of 1-3 falls in the previous six months will participate in Cranial Nerve Non-Invasive Neuromodulation enhanced gait and balance training.
  Interventions: Device: Cranial Nerve Non-Invasive Neuromodulation
- Young Adult - Control (Active Comparator): Healthy subjects between the ages of 18-39 will participate in Sham Cranial Nerve Non-Invasive Neuromodulation gait and balance training.
  Interventions: Behavioral: Sham Cranial Nerve Non-Invasive Neuromodulation

INTERVENTIONS:
Device: Cranial Nerve Non-Invasive Neuromodulation — Portable device delivers electrical stimulation to cranial nerves V and VII via an electrode array placed on the anterior surface of the tongue. Stimulation is combined with rehabilitation exercises targeting walking and balance.
  Other Names: PoNS (Portable Neuromodulation Stimulator)
  Arms: Healthy Older Adults - Intervention; Older Fallers - Intervention; Young Adults - Intervention
Behavioral: Sham Cranial Nerve Non-Invasive Neuromodulation — Subjects participate in gait and balance rehabilitation exercises while using a device set to sub-threshold levels.
  Arms: Healthy Older Adults - Control; Older Fallers - Control; Young Adult - Control

SUMMARY:
The purpose of this study is twofold:

1. Establish baseline measures of gait performance in healthy young and older adults, and older adults with a history of falls.
2. Investigate the effects of gait and balance training with and without cranial nerve noninvasive neuromodulation (CN-NINM) on postural balance and gait performance in older adults.

For the second purpose, the study will incorporate a placebo-controlled design to evaluate the effects of CN-NINM augmented exercise compared to physical exercises alone. Both groups will perform gait and postural balance training (outlined in more detail below) but will differ in the stimulation level of the PoNS device. The investigators will use the results of this study as a first step toward evaluating the benefits of CN-NINM in a falls prevention program.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling
* Able to understand and give informed consent
* Able to stand and walk independently without an assistive device
* No contraindication to exercise

  1. Healthy young adults
* Between ages of 18 and 39
* Scores above 19 on Dynamic Gait Index 2. Healthy older adults without a history of falls
* Age 65+
* Scores above 19 on Dynamic Gait Index 3. Older adults with a history of falls
* Age 65+
* Self-reported history of 1-3 falls in previous year
* Scores of 19 and below on the Dynamic Gait Index

Exclusion Criteria:

* History of musculoskeletal disorders (lower-limb joint replacement, radiographic evidence of severe osteoarthritis, broken leg bone or ligament/tendon injury in prior 6 months)
* Use of tobacco products
* Any oral abrasions, cuts, cold sores, piercings, tissue inflammation, or have had oral surgery within the previous 3 months
* Have a pacemaker or are identified as at-risk for cardiovascular events
* Have a biomechanical prosthetic
* If female, self-report of being pregnant
* Neurological condition
* Prisoners
* Individuals clearly lacking the capacity to provide informed consent

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2013-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Dynamic Gait Index | Day 1 and approximately Day 12
  An 8-item inventory of functional gait tasks each scored on a 0-3 point scale. Maximum score is 24 and any score of 19 or lower indicates an increased risk of falling.

CONTACTS AND LOCATIONS:
Overall Officials: Darryl G Thelen, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States